CLINICAL TRIAL: NCT05865847
Title: Unveiling the Alcohol Harm Paradox: Analysis of Socioeconomic Differences in Alcohol Harm in Finland in a Nationwide Cohort Study
Brief Title: Socioeconomic Differences in Alcohol Harm in Finland in a Nationwide Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Social Insurance Institution, Finland (Other)
Responsible Party: Sponsor
Other Study IDs: KKO-Inv 4-Johto-VPT-Terveysind
Record Dates: First submitted 2023-05-03; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Alcohol-Related Disorders
MeSH Terms: conditions — Alcohol-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lowest income groups: Deciles of equivalized net household income. The method compares the whole socioeconomic distribution.
  Interventions: Other: Not applicable, this is an observational study

INTERVENTIONS:
Other: Not applicable, this is an observational study — Not applicable, this is an observational study

SUMMARY:
This is a nationwide cohort study of Finnish adults aged 25 and older, who are followed up for the incidence of an alcohol-attributable hospitalization or death. The primary objective is to examine the relative and absolute socioeconomic differences in cause-specific alcohol-attributable hospital admissions and deaths.

DETAILED DESCRIPTION:
Background

Alcohol consumption is a leading risk factor for death and disability, resulting in substantial societal costs and social and community harm. Alcohol-related harm has been consistently shown to be higher among people of lower socioeconomic status, despite the fact they often report similar or lower levels of alcohol use. This apparent contrast has been called the alcohol harm paradox.

Understanding what explains the alcohol harm paradox is crucial for the design and implementation of population health interventions to reduce socioeconomic differences in alcohol harm. Explanations for the paradox can be broadly categorised into three groups: (i) differential exposure to alcohol, drinking patterns and trajectories and to other behavioural risk factors and joint effects among them, (ii) differential vulnerability resulting from individual factors, such as biological characteristics, psychological traits or stress, cumulative disadvantage and broader community and societal upstream factors, and (iii) differential biases in the measurement of alcohol exposure.

A crucial weakness of existing empirical studies comes from the operationalization of alcohol harm. With few exceptions, a vast majority of studies has used a composite endpoint combining several causes of alcohol-attributable deaths or hospitalizations or even merging alcohol-attributable hospital admissions with deaths in a single outcome. While this strategy increases the statistical power to analyse rare events, composite endpoints are prone to misclassification bias by masking divergent underlying patterns and associations.

Cause-specific analyses might shed light on different mechanisms driving the socioeconomic differences in overall alcohol-attributable harm, as well as opening potential avenues for policy interventions to reduce them. The study will take advantage of a recently formed dataset covering the total Finnish population to explore associations between socioeconomic status and cause-specific alcohol-attributable events. An additional contribution to the literature will be reporting both relative and absolute inequalities in alcohol-attributable harm. Absolute differences have been rarely reported even though might be as relevant as relative differences because, from a pragmatic standpoint, they are more feasible to reduce.

The study will aim to (1) examine the relative and absolute socioeconomic differences in cause-specific alcohol-attributable hospital admissions and deaths; (2) describe the geographical differences in cause-specific alcohol-attributable hospital admissions and deaths; and (3) quantify the relative contribution of each specific alcohol-attributable cause to the overall alcohol-attributable harm.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents (defined by Statistics Finland as those Finnish and foreign nationals who have a legal domicile in Finland and intend to stay (or have stayed) for at least one year) alive in Finland by December 31, 2015
* Age 25 years or older by January 1, 2016
* Not having an alcohol-attributable hospitalization during the past three years ((January 2013-December 2015

Exclusion Criteria:

* Temporary residents, including foreign nationals living in Finland for less than a year, asylum seekers who have not been granted a legal domicile, temporary migrant workers and Finnish nationals living temporarily abroad by December 31, 2015

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All permanent residents in Finland older than 25 years old and without an alcohol-attributable hospital admission during the past three years
Sampling Method: Probability Sample
Enrollment: 3950000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol intoxication - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of alcohol intoxication hospitalization (ICD-10 F10.0-1)
Alcohol intoxication - Death | January 1, 2016 to February 28, 2020
  Death due to alcohol intoxication (ICD-10 F10.0-1)
Alcohol dependence - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of hospitalization due to alcohol dependence (F10.2)
Alcohol dependence - Death | January 1, 2016 to February 28, 2020
  Death due to alcohol dependence (F10.2)
Psycho-organic syndrome caused by alcohol - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of hospitalization due to psycho-organic syndrome caused by alcohol (F10.3-9)
Psycho-organic syndrome caused by alcohol - Death | January 1, 2016 to February 28, 2020
  Death due to psycho-organic syndrome caused by alcohol (F10.3-9)
Alcoholic liver disease - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of hospitalization due to alcoholic liver disease(K70)
Alcoholic liver disease - Death | January 1, 2016 to February 28, 2020
  Death due to alcoholic liver disease(K70)
Pancreatic diseases caused by alcohol - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of hospitalization due to pancreatic diseases caused by alcohol (K85.2, K86.0)
Pancreatic diseases caused by alcohol - Death | January 1, 2016 to February 28, 2020
  Death due to pancreatic diseases caused by alcohol (K85.2, K86.0)
Gastritis caused by alcohol - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of hospitalization due to gastritis caused by alcohol (K29.2)
Gastritis caused by alcohol - Death | January 1, 2016 to February 28, 2020
  Death due to gastritis caused by alcohol (K29.2)
Alcoholic cardiomyopathy - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of hospitalization due to alcoholic cardiomyopathy (I42.6)
Alcoholic cardiomyopathy - Death | January 1, 2016 to February 28, 2020
  Death due to alcoholic cardiomyopathy (I42.6)
Nervous system disorders caused by alcohol - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of hospitalization due to degeneration of the nervous system due to alcohol, epileptic seizures related to alcohol, alcoholic polyneuropathy, alcoholic myopathy (G312, G4051, G621, G721)
Nervous system disorders caused by alcohol - Death | January 1, 2016 to February 28, 2020
  Death due to degeneration of the nervous system due to alcohol, epileptic seizures related to alcohol, alcoholic polyneuropathy, alcoholic myopathy (G312, G4051, G621, G721)
Alcohol poisoning - Hospitalization | January 1, 2016 to February 28, 2020
  Incidence of hospitalization due to alcohol poisoning (T51, X45)
Alcohol poisoning - Death | January 1, 2016 to February 28, 2020
  Death due to alcohol poisoning (T51, X45)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Peña, MD, PhD, Principal Investigator — Finnish Institute for Health and Welfare; Sonja Lumme, PhD, Study Chair — Finnish Institute for Health and Welfare; Päivikki Koponen, PhD, Study Chair — Finnish Institute for Health and Welfare

IPD SHARING:
Plan to Share IPD: No
The investigators will share the harmonization protocol to define the variables and the statistical code. Individual participant data is available upon request at FinData, following national data protection procedures.

REFERENCES:
- [Background] GBD 2016 Alcohol Collaborators. Alcohol use and burden for 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2018 Sep 22;392(10152):1015-1035. doi: 10.1016/S0140-6736(18)31310-2. Epub 2018 Aug 23. PMID 30146330
- [Background] Manthey J, Hassan SA, Carr S, Kilian C, Kuitunen-Paul S, Rehm J. What are the Economic Costs to Society Attributable to Alcohol Use? A Systematic Review and Modelling Study. Pharmacoeconomics. 2021 Jul;39(7):809-822. doi: 10.1007/s40273-021-01031-8. Epub 2021 May 10. PMID 33970445
- [Background] Room R, Ferris J, Laslett AM, Livingston M, Mugavin J, Wilkinson C. The drinker's effect on the social environment: a conceptual framework for studying alcohol's harm to others. Int J Environ Res Public Health. 2010 Apr;7(4):1855-71. doi: 10.3390/ijerph7041855. Epub 2010 Apr 21. PMID 20617064
- [Background] Probst C, Lange S, Kilian C, Saul C, Rehm J. The dose-response relationship between socioeconomic deprivation and alcohol-attributable mortality risk-a systematic review and meta-analysis. BMC Med. 2021 Nov 5;19(1):268. doi: 10.1186/s12916-021-02132-z. PMID 34736475
- [Background] Probst C, Kilian C, Sanchez S, Lange S, Rehm J. The role of alcohol use and drinking patterns in socioeconomic inequalities in mortality: a systematic review. Lancet Public Health. 2020 Jun;5(6):e324-e332. doi: 10.1016/S2468-2667(20)30052-9. PMID 32504585
- [Background] Syden L, Sidorchuk A, Makela P, Landberg J. The contribution of alcohol use and other behavioural, material and social factors to socio-economic differences in alcohol-related disorders in a Swedish cohort. Addiction. 2017 Nov;112(11):1920-1930. doi: 10.1111/add.13889. Epub 2017 Jul 17. PMID 28556302
- [Background] Makela P, Paljarvi T. Do consequences of a given pattern of drinking vary by socioeconomic status? A mortality and hospitalisation follow-up for alcohol-related causes of the Finnish Drinking Habits Surveys. J Epidemiol Community Health. 2008 Aug;62(8):728-33. doi: 10.1136/jech.2007.065672. PMID 18621959
- [Background] Pena S, Makela P, Laatikainen T, Harkanen T, Mannisto S, Heliovaara M, Koskinen S. Joint effects of alcohol use, smoking and body mass index as an explanation for the alcohol harm paradox: causal mediation analysis of eight cohort studies. Addiction. 2021 Aug;116(8):2220-2230. doi: 10.1111/add.15395. Epub 2021 Jan 28. PMID 33404149
- [Background] Katikireddi SV, Whitley E, Lewsey J, Gray L, Leyland AH. Socioeconomic status as an effect modifier of alcohol consumption and harm: analysis of linked cohort data. Lancet Public Health. 2017 May 10;2(6):e267-e276. doi: 10.1016/S2468-2667(17)30078-6. eCollection 2017 Jun. PMID 28626829
- [Background] Makela P. Alcohol-related mortality as a function of socio-economic status. Addiction. 1999 Jun;94(6):867-86. doi: 10.1046/j.1360-0443.1999.94686710.x. PMID 10665076
- [Background] Pena S, Makela P, Harkanen T, Heliovaara M, Gunnar T, Mannisto S, Laatikainen T, Vartiainen E, Koskinen S. Measurement error as an explanation for the alcohol harm paradox: analysis of eight cohort studies. Int J Epidemiol. 2021 Jan 23;49(6):1836-1846. doi: 10.1093/ije/dyaa113. PMID 32995840
- [Background] Sadler S, Angus C, Gavens L, Gillespie D, Holmes J, Hamilton J, Brennan A, Meier P. Understanding the alcohol harm paradox: an analysis of sex- and condition-specific hospital admissions by socio-economic group for alcohol-associated conditions in England. Addiction. 2017 May;112(5):808-817. doi: 10.1111/add.13726. Epub 2017 Feb 6. PMID 27981670
- [Background] Mackenbach JP, Kulhanova I, Bopp M, Borrell C, Deboosere P, Kovacs K, Looman CW, Leinsalu M, Makela P, Martikainen P, Menvielle G, Rodriguez-Sanz M, Rychtarikova J, de Gelder R. Inequalities in Alcohol-Related Mortality in 17 European Countries: A Retrospective Analysis of Mortality Registers. PLoS Med. 2015 Dec 1;12(12):e1001909. doi: 10.1371/journal.pmed.1001909. eCollection 2015 Dec. PMID 26625134
- [Background] Mackenbach JP. Should we aim to reduce relative or absolute inequalities in mortality? Eur J Public Health. 2015 Apr;25(2):185. doi: 10.1093/eurpub/cku217. No abstract available. PMID 25818489

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT05865847/Prot_SAP_000.pdf